CLINICAL TRIAL: NCT04246710
Title: Pancreatic Cancer Molecular Sub-classification for Prognostic Stratification and Individualized Therapy Using Endoscopic Ultrasound Tissue Core Biopsy Samples
Brief Title: Pancreatic Cancer Molecular Sub-classification Using Endoscopic Ultrasound Tissue Core Biopsy Samples
Status: Active, not recruiting | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Guido Costamagna, Professor, Catholic University of the Sacred Heart
Other Study IDs: PDAC-SUBCLASS
Record Dates: First submitted 2020-01-19; First posted 2020-01-29 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Pancreas Cancer
Keywords: pancreatic cancer; EUS; molecular subtyping; personalized medicine
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — sequencing on DNA from paraffin tissues will be performed to examine the mutational and copy number status of 87 genes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluated the feasibility and reliability of PDAC molecular subtyping on tissue core biopsies samples acquired under EUS guidance. Moreover, this study will assess the impact of molecular subtypes assessed on EUS-FNB samples in patients with resectable and unresectable (locally advanced, advanced, and metastatic) PDAC undergoing chemotherapy on treatment response and survival and the utility in monitoring disease response to therapy and early occurrence of disease relapse using the TaqMan RNA assay in serum

DETAILED DESCRIPTION:
PDAC patients are categorised as resectable, borderline resectable, locally advanced, metastatic and recurrent. Substantial neoplastic tissue is only available for the resectable group. This is unfortunate as the other groups are those that would benefit the most from molecular characterization and identification of markers, which may be predictive and/or provide therapeutic stratification. For these categories of patients, only fine needle aspiration or small biopsies could be obtained until now. However, the introduction of new needles, specifically designed to acquire larger high quality biopsy samples under endoscopic ultrasound (EUS), has now made it possible to test prognostic, predictive and therapeutic stratification markers. However, the applicability of EUS-fine needle biopsy (EUS-FNB) samples for this purpose has yet to be clinically validated. The working hypothesis of this proposal is that the molecular sub-classification of PDAC on EUS-FNB tissue samples could be applied for prognostic stratification and therapeutic decision strategies in both resectable and unresectable patients using DNA and RNA biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to EUS with FNB in the suspect of pancreatic cancer
* Availability of biopsies obtained during EUS-FNB
* Histological diagnosis of pancreatic ductal adenocarcinoma of any stage
* Age >18 and <80 years
* Willing to be followed up at the Fondazione Policlinico A. Gemelli University Hospital
* Able to sign informed consent

Exclusion Criteria:

* Histological diagnoses other than pancreatic ductal adenocarcinoma
* Pregnancy or lactation
* Unable to sigh informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study concerns consecutive individuals with a solid pancreatic lesion who will undergo diagnostic EUS-FNB. Those with a histological diagnosis of PDAC will be enrolled in the study. Enrollment will include patients with resectable disease and those with unresectable disease, which can be divided in different stages, i.e. borderline resectable, locally advanced, advanced, and metastatic.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2018-01-28 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility of PDAC molecular subtyping on biopsy samples | At 6 months
  Number of patients in whom molecular subtyping on biopsy samples is obtained
Reliability of PDAC molecular subtyping on biopsy samples | At 1 year
  concordance between molecular subtyping on biopsy samples and surgery specimens

SECONDARY OUTCOMES:
Progression-free-survival (PFS) | From date of enrollment assessed until death or up to 3 years
  To assess the impact of molecular subtypes assessed on EUS-FNB samples PFS defined as the time from the date of trial entry until disease progression or relapse.
Overall survival | From date of enrollment assessed until death or up to 3 years
  Overall survival defined as the length of time (in days) between the treatment date and the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Larghi, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli
Locations (1):
- Universita' Cattolica del Sacro Cuore, Rome, Italy

IPD SHARING:
Plan to Share IPD: No